CLINICAL TRIAL: NCT02545140
Title: Prevention Strategies for Adolescents at Risk of Diabetes - Validation of a Risk Tool for Young People Aged 12 - 14 Years
Brief Title: Prevention Strategies for Adolescents at Risk of Diabetes
Acronym: PRE-STARt
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Collaborators: University of Leicester (Other); Associacao Protectora dos Diabeticos de Portugal (Other); The Algarve Regional Health Administration (Other); University of Leipzig (Other); Technische Universität Dresden (Other); Alexander Technological Educational Institute, Thessaloniki, Greece (Other); Diabetes Centre of Paediatrics P&A (Unknown); Athens General Children's Hospital "Pan. & Aglaia Kyriakou" (Other); Primary Care Centre Egia, San Sebastian, Spain (Unknown); Basque Government Department of Public Health (Other); Health Department of the Alto/Bajo Deba (Other)
Responsible Party: Sponsor
Other Study IDs: 173431
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes; Chronic Disease
Keywords: risk factors; screening; adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- UK (Lead Site): Data will be collected from 100 adolescents from each participating site providing clinical data for 500 adolescents providing a cross-sectional cohort from each of the following countries:
  UK (Lead Site) Germany Portugal Greece Spain (Basque Country)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The primary aim of PRE-STARt Phase 1 is to pragmatically evaluate and refine a risk assessment tool to identify those children with chronic disease risk factors (including Type 2 Diabetes).

DETAILED DESCRIPTION:
Data will be collected in 5 European Commission countries (500 adolescents in total). A range of biological and lifestyle measures will be collected in order to investigate the adolescent's lifestyle and will include body weight and other anthropometric measurements, blood pressure, blood capillary sample, self-reported physical activity, sedentary behaviour and dietary habits. Their parent/guardian will complete a number of questions to gather information about variables that have been associated with chronic disease (including type 2 diabetes) and include peri-natal history (birth weight, gestational diabetes), socioeconomic status, family health and medical history.

A draft risk tool to identify those children with a 'higher risk' of developing type 2 diabetes in the future has been developed systematic review results and a Delphi procedure. This draft tool will be evaluated and refined. This draft risk tool will be evaluated by independent clinical reviewers against the data collected from the 500 adolescent data sets. The results for each adolescent will be independently reviewed by clinicians who will assign either a "lower" or "higher" risk to each case. The results will be compared to the results from the draft 'PRE-START tool', used to further refine this identification tool using appropriate statistical methods.

The outputs of this study will be a fit for purpose 'PRE-STARt tool' that can be used for recruitment to interventional studies whose primary objective is to reduce the risk of developing chronic disease (including type 2 diabetes) in the future.

ELIGIBILITY:
Inclusion Criteria:

* Young people aged between 12-14 years of age
* be willing and able to give assent
* have obtained written parent/guardian consent.

Exclusion Criteria:

* are outside the age range of interest (i.e. aged less than 12 years or greater than 14 years of age)
* do not have parental consent or do not give assent
* have an existing diagnosis of type 1 or type 2 diabetes

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Boys and girls who are between 12 and 14 years of age who do not have an existing diagnosis of type 1 or type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Chronic disease risk factor - Body mass index (BMI) | 12 months
  Height and weight will be measured to calculated BMI

SECONDARY OUTCOMES:
Chronic disease risk factor - waist circumference | 12 months
Chronic disease risk factor - blood pressure | 12 months
Chronic disease risk factor - glycated haemoglobin (HbA1c) | 12 months
Chronic disease risk factor - high density lipoprotein cholesterol | 12 months
Chronic disease risk factor - glucose | 12 months
  Fasted and/or unfasted
Chronic disease risk factor - low density lipoprotein cholesterol | 12 months
  Calculated
Chronic disease risk factor - triglycerides | 12 months
Chronic disease risk factor - total cholesterol | 12 months

OTHER OUTCOMES:
Risk tool refinement | 18 months
  A draft risk tool to identify those children with a 'higher risk' of developing type 2 diabetes in the future that has been developed systematic review results and a Delphi procedure. Each adolescent will complete a diet and lifestyle questionnaire about their physical activity, sedentary behaviour and dietary habits and the parent/guardian will complete a questionnaire about their family health history and about their child's early years (including gestational period, birth weight, whether they were breast or bottle fed). This draft tool will be evaluated and refined using these data and the data from the assessments mentioned in 1-9. The draft risk tool will then be refined based on data from the 500 adolescents using appropriate statistical methods resulting in an externally validated risk tool that can be used to screen young people aged between 12-14 years for being at risk of developing of type 2 diabetes in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Davies, MD, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, United Kingdom